CLINICAL TRIAL: NCT05353829
Title: Efficacy, Tolerability and Preferences of Per Oral or Subcutaneous Methotrexate in Patients with Early Rheumatoid Arthritis - a Randomised Register Based Multicentre Study
Brief Title: Methotrexate in Patients with Early Rheumatoid Arthritis
Acronym: MTXRA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Region Västerbotten (Other Government)
Collaborators: Region Gävleborg (Other); Umeå University (Other); Uppsala University (Other); County Council of Norrbotten, Sweden (Other Government); Vastra Gotaland Region (Other Government); Västernorrland County Council, Sweden (Other Government); Dalarna County Council, Sweden (Other); Karolinska University Hospital (Other); Region Jämtland Härjedalen (Other); Sormland County Council, Sweden (Other); Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Anna Södergren, Principal Investigator, Region Västerbotten
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTXRA; 2020-000462-41 (EudraCT Number)
Record Dates: First submitted 2021-05-11; First posted 2022-04-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arhtritis; methotrexate; registerbased randomisation; health economics; patient preferences; gut microbiota
MeSH Terms: conditions — Arthritis, Rheumatoid; Patient Preference | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Per oral (Active Comparator): Drug:per oral Methotrexate Tablets dosage 5-30mg once weekly.
  Interventions: Drug: Methotrexate
- Subcutaneous (Active Comparator): Drug: subcutaneous Methotrexate Injection dosage 5-30mg once weekly.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — When accepted inclusion the patient will be included in SRQ, and thereafter randomised for Methotrexate per oral or subcutaneous administration

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease primarily affecting the small joints of hands and feet, but may also present with systemic, extraarticular features. The Swedish Rheumatology Quality Register (SRQ) is a nationwide quality register with the aim of continuously improving the treatment and follow-up of patients with rheumatic disease. Using this type of quality registers, it is possible to perform a Registrybased Randomised Clinical Trial (R-RCT), that is a randomised clinical trial this is carried out by screening, recruitment and registration of study data is performed based on information given by a quality register. All patients with newly diagnosed RA are included in SRQ. Treatment options for RA include different types of immunosuppression and corticosteroids as bridging therapy. Methotrexate, a synthetic conventional disease modifying antirheumatic drug (csDMARD), which can be given either orally or subcutaneously, is considered a first-line treatment. Studies have shown the beneficial efficacy and improved quality of life for patients with RA treated with methotrexate, however this is not studied in a setting of unselected patients with newly diagnosed RA in northern Sweden. Moreover, it is not known to what extent patients prefer oral or subcutaneous administration route, or if there are any health economic benefits from either of the two administration routes. Further, changes in gut microbiota is not studied in this setting.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic inflammatory disease primarily affecting the small joints of hands and feet, but may also present with systemic, extraarticular features. Pain and stiffness induced by rest, fever, fatigue, and weight loss are common constitutional symptoms. After onset of symptoms the patient most often sees a general practitioner for referral to a rheumatology department. After diagnosis of RA treatment is indicated to start as soon as possible to prevent future disability. Treatment options for RA include different types of immunosuppression and corticosteroids as bridging therapy. Methotrexate (MTX) has been used for decades as the most commonly prescribed synthetic conventional disease modifying antirheumatic drug (csDMARD) in the treatment for RA. MTX can be given either orally or subcutaneously, although the most commonly used route is still per oral, largely due to convenience. Studies have shown the beneficial efficacy and improved quality of life with methotrexate treatment. Although its mechanism of action has not been fully elucidated, current evidence supports that it works by acting as both an antimetabolite (by inhibiting dihydrofolate reductase) and an immunomodulatory agent (by promoting adenosine release, thereby suppressing inflammation). MTX has long been used as a standard of care to treat RA at typically between 7.5 and 30.0 mg/week in a single weekly dose. Methotrexate has a broad spectrum of adverse effects, one of which is the most common is gastrointestinal manifestations. In our clinic, the standard clinical practice is to start with per oral administration and then a switch from oral medication to subcutaneous injections in cases where gastrointestinal adverse effects occur or a failure to reach remission. When given subcutaneously, the bioavailability of methotrexate increases which thereby is thought to enhance the efficacy of methotrexate. A recent metanalysis showed that subcutaneously given MTX therapy has significantly higher odds than single dose weekly oral MTX of achieving reduction in disease activity, with no increased adverse effects. However, this metanalysis also pinpoints the fact that studies in this area is surprisingly few, i.e. this metanalysis is only based on four original publications.

The Swedish Rheumatology Quality Register (SRQ) is a nationwide quality register with the aim of continuously improving the treatment and follow-up of patients with rheumatic disease. SRQ has been granted certification level

1, which is the highest level a national quality register can obtain. Using this type of quality registers, it is possible to perform a Registrybased Randomised Clinical Trial (R-RCT) that are defined as prospective randomised studies that to some extent use registers for their implementation, that is for example a randomised clinical trial carried out by screening, recruitment and registration of study data based on information given in a quality register. Studies have also proposed an effect on gut microbiota both by the RA disease itself as well as by treatment with methotrexate. There is increasing knowledge that the gut microbiota are not only involved in the digestion and absorption of food, but they can also exert a protective function by preventing adherence of pathogenic bacteria to the mucosal layer, and they play a pivotal role in modulating the innate and acquired immunity of the host. Remarkably, gut microbiota exert their effects not only in the intestine but can signal to distant organs in the body, thereby explaining their association with several diseases, including RA. From a clinical perspective, elucidation of the interaction between RA, MTX and the gut microbiota could reduce the costs and harm to patients that is caused by "trial and error" use of drugs with highly variable treatment responses. Patient acceptability is particularly significant in dictating adherence to therapy.

A potential drawback to subcutaneous MTX is patients' fear of needles and/ or the discomfort of selfinjecting; however, this doubt has been strongly reassured with the advent of the widely accepted biologics which require self-injection. Recent studies examined patient preferences for RA treatment in several populations, finding that most participants were willing to accept certain risks of adverse effects to gain potential benefits, however there seem to be a variability in patient preferences for RA treatment, highlighting the importance of incorporating patient input into the treatment approach. Previous studies have mainly focused on patients with established RA, showing that many patients place a high value on treatment benefits over other treatment attributes, including side effects, cost, or route of administration (9) and also an expectance for injections of MTX in patients with long standing RA. However, patient preference studies are scarce in patients with newly diagnosed disease and in our part of the world. For patient preference study a (threshold technique) TT exercise is often used. Here a decisionmaker, typically a patient or physician is presented with a choice between two treatment or healthcare delivery options. One is the reference option that is the baseline against which an alternative is compared. It is often the option associated with the status quo or standard of care. The second is the target option and confers both an incremental benefit and an incremental burden relative to the status quo or standard of care. Once the reference and target options have been identified, the researcher must identify the key attribute of the target option (either a benefit or a burden) that will be used to estimate the strength of preference for the target relative to the reference option. The key attribute can be any attribute for which values can be expressed numerically. The most common key attributes are probability of benefit, risk of harm, waiting time, life expectancy, and cost. When the key attribute is a measure of burden (e.g., risk of harm, waiting time, or cost), the estimated threshold is a measure of the additional burden that exactly offsets the incremental benefit of the target option. If the key attribute is a benefit (e.g., probability of benefit or life expectancy), the estimated threshold is a measure of the minimum additional benefit that the target must provide to offset the incremental burden of that option. After being presented with descriptions of the two options, respondents real-world options with well-known attributes, using all available information in the initial question, including known differences between the options in the value of the key attribute, may provide a direct measure of decision makers' preference between the reference and target options in addition to providing a starting point for estimating the threshold value of the key attribute. If the reference option is chosen in the initial question, the key attribute of the target is made better or more appealing and the question is repeated. If the target is chosen initially, the key attribute of the target is made worse or less appealing and the question is repeated. The process continues until the researcher can identify the threshold level of the key attribute, i.e., the level at which a respondent is indifferent between the reference and target options. The difference between the threshold value of the key attribute and the level of the same attribute in the reference option is a measure of the strength of preference for the target option compared with the reference option. It is a measure of the change in the key attribute that exactly offsets the difference in benefit or burden between the reference and the target options. The threshold can be a specific value or an interval within which the threshold lies. If the tradeoff exercise yields a specific value, then that threshold for each respondent for each trade-off exercise is known. If, however, the trade-off exercise results in a threshold interval, then the researcher has options for how to utilize these data. The researcher can simply report the threshold interval or the proportion of respondents choosing the target option at different threshold intervals. During recent year an increasing interest have been on cost-utility analyses, comparing the cost per quality-adjusted life-year (QALY) of different treatment regimes. However, most studies focus on biologic treatment. The incremental cost for subcutaneous compared to per oral methotrexate is not insignificant, still health economic evaluations comparing these two administration routes, and which administration to recommend, are scarce.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written consent to participate in the study
* Diagnosis of rheumatoid arthritis by rheumatologist fulfilling 2010
* Rheumatoid Arthritis Classification Criteria
* Indication of methotrexate
* 18-95 years of age
* Women of Childbearing Capacity (WOCBC) must:

  1. Comply to use of highly effective contraception methods during the course of the trial.
  2. Have a negative pregnancy test.
* Male patients included in the study that have fertile female partners must use adequate contraception within their relationship during the same period of time

Exclusion Criteria:

* Contraindications for methotrexate
* Previous treatment with any DMARD within the last five years
* Known or suspected allergies against methotrexate or any other substance in the given medication
* Anamnestic information on pregnancy, breastfeeding, or planned pregnancy
* Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation or inability to answer questionnaire in written Swedish
* Treatment or disease which, according to the investigator, can affect treatment or study results.
* Fear of needles leading to not being able to use subcutaneous injections
* For the study in gut microbiota: Use of antibiotics or probiotics within the last 3 months

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease activity measured as DAS28 over 12 months | 12 months
  The primary objective of this study is to study difference in DAS28 (range 0-10, higher value means higher disease activity) over 12 months of follow up in patients with newly diagnosed RA randomized to oral or subcutaneous methotrexate

SECONDARY OUTCOMES:
Disease activity measured as DAS28 over 24 months | 24 months
  One secondary outcome is to study difference disease activity measured as DAS28 (range 0-10, higher value means higher disease activity) over 24 months of follow up in patients with newly diagnosed RA randomized to oral or subcutaneous methotrexate
Disease activity measured as DAS28 over 3 months | 3 months
  One secondary outcome is to study difference disease activity measured as DAS28 (range 0-10, higher value means higher disease activity) over 3 months of follow up in patients with newly diagnosed RA randomized to oral or subcutaneous methotrexate
Disease activity measured as DAS28 over 6 months | 6 months
  One secondary outcome is to study difference disease activity measured as DAS28 (range 0-10, higher value means higher disease activity) over 6 months of follow up in patients with newly diagnosed RA randomized to oral or subcutaneous methotrexate
Gut microbiota by sequencing of the microbial 16S rRNA gene | 24 months
  At follow up nalysis of gut microbiota composition will be done by sequencing of the microbial 16S rRNA gene.
Patient preferences | 24 months
  To determine the acceptable levels of risks for newly diagnosed patients with RA measured using the threshold technique
Health economy | 24 months
  To determine the health economic aspects including quality of life, measured by EQ5D, of the two administration routes
Adverse events | 24 months
  Number of adverse events in patients with newly diagnosed RA randomized to oral or subcutaneous methotrexate over 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Anna Södergren, MD PhD, Principal Investigator — Region Västerbotten
Locations (13):
- Sweden (13):
  - Region Sörmland, Eskilstuna
  - Region Dalarna, Falun
  - Region Gävleborg, Gävle
  - Region Norrbotten, Luleå
  - Reumatologsektionen Örebro universitetssjukhus, Öre
  - Region Jämtland Härjedalen, Östersund
  - Västra Götalandsregionen, Skövde
  - Akademiskt specialistcentrum, Stockholm
  - Danderyds sjukhus, Stockholm
  - Karolinska sjukhuset, Stockholm
  - Region Västernorrland, Sundsvall
  - Region Västerbotten, Umeå
  - Reumatologisk klinik, Västerås, Västerås

IPD SHARING:
Plan to Share IPD: No
Individual level data may not be made publicly available due to The General Data Protection Regulation (GDPR) and privacy concerns. The data used for this study contain protected health information. Data will available from Umeå University for researchers who meet the criteria for access to confidential data and have entered into a data use agreement. Umeå University has restricted public sharing because they contain identifying patient information.

REFERENCES:
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Visser K, van der Heijde D. Optimal dosage and route of administration of methotrexate in rheumatoid arthritis: a systematic review of the literature. Ann Rheum Dis. 2009 Jul;68(7):1094-9. doi: 10.1136/ard.2008.092668. Epub 2008 Nov 25. PMID 19033290
- [Background] Schiff M, Weinblatt ME, Valente R, van der Heijde D, Citera G, Elegbe A, Maldonado M, Fleischmann R. Head-to-head comparison of subcutaneous abatacept versus adalimumab for rheumatoid arthritis: two-year efficacy and safety findings from AMPLE trial. Ann Rheum Dis. 2014 Jan;73(1):86-94. doi: 10.1136/annrheumdis-2013-203843. Epub 2013 Aug 20. PMID 23962455
- [Background] Bujor AM, Janjua S, LaValley MP, Duran J, Braun J, Felson DT. Comparison of oral versus parenteral methotrexate in the treatment of rheumatoid arthritis: A meta-analysis. PLoS One. 2019 Sep 6;14(9):e0221823. doi: 10.1371/journal.pone.0221823. eCollection 2019. PMID 31490947
- [Background] Picchianti-Diamanti A, Panebianco C, Salemi S, Sorgi ML, Di Rosa R, Tropea A, Sgrulletti M, Salerno G, Terracciano F, D'Amelio R, Lagana B, Pazienza V. Analysis of Gut Microbiota in Rheumatoid Arthritis Patients: Disease-Related Dysbiosis and Modifications Induced by Etanercept. Int J Mol Sci. 2018 Sep 27;19(10):2938. doi: 10.3390/ijms19102938. PMID 30261687
- [Background] Sayers E, MacGregor A, Carding SR. Drug-microbiota interactions and treatment response: Relevance to rheumatoid arthritis. AIMS Microbiol. 2018 Oct 26;4(4):642-654. doi: 10.3934/microbiol.2018.4.642. eCollection 2018. PMID 31294239
- [Background] Schroeder BO, Backhed F. Signals from the gut microbiota to distant organs in physiology and disease. Nat Med. 2016 Oct;22(10):1079-1089. doi: 10.1038/nm.4185. Epub 2016 Oct 6. PMID 27711063
- [Background] Hsiao B, Fraenkel L. Patient preferences for rheumatoid arthritis treatment. Curr Opin Rheumatol. 2019 May;31(3):256-263. doi: 10.1097/BOR.0000000000000591. PMID 30747733
- [Background] Durand C, Eldoma M, Marshall DA, Bansback N, Hazlewood GS. Patient Preferences for Disease-modifying Antirheumatic Drug Treatment in Rheumatoid Arthritis: A Systematic Review. J Rheumatol. 2020 Feb;47(2):176-187. doi: 10.3899/jrheum.181165. Epub 2019 Apr 15. PMID 30988125
- [Background] Striesow F, Brandt A. Preference, satisfaction and usability of subcutaneously administered methotrexate for rheumatoid arthritis or psoriatic arthritis: results of a postmarketing surveillance study with a high-concentration formulation. Ther Adv Musculoskelet Dis. 2012 Feb;4(1):3-9. doi: 10.1177/1759720X11431004. PMID 22870490